CLINICAL TRIAL: NCT03448445
Title: An Observational Study to Evaluate AD Conversion Rate Differences Between High-risk MCI and Low Risk MCI in Real World Setting
Brief Title: A Study to Evaluate Alzheimer's Disease Conversion Rate Differences Between High-risk Mild Cognitive Impairment (MCI) and Low-risk MCI in a Real World Setting
Acronym: CONCORDE
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E0000-M082-603
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-05

CONDITIONS: Mild Cognitive Impairment
Keywords: High-risk; Low-risk; Alzheimer's disease; Observational study
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk MCI: This cohort will include participants with high-risk mild cognitive impairment (MCI).
  Interventions: Other: Usual care setting
- Low-risk MCI: This cohort will include participants with low-risk MCI.
  Interventions: Other: Usual care setting

INTERVENTIONS:
Other: Usual care setting — usual care settings without any intervention

SUMMARY:
This study will be conducted to evaluate the rate of Alzheimer's disease conversion differences between high-risk mild cognitive impairment (MCI) and low-risk MCI.

ELIGIBILITY:
Inclusion Criteria:

* Participant over 55 years old and less than 90 years old
* Participant with subjective memory complaint by informant
* Clinical Dementia Rating (CDR) of 0.5; memory score box must be at least 0.5
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease cannot be made by the site physician at the time of the screening visit
* Essentially preserved activities of daily living
* Absence of dementia
* Participant with Seoul Neuropsychological Screening Battery-Dementia Version cut-off score between 134.25 and 188.25
* Participants and caregivers who give written authorization to use their personal and health data
* Cognitive decline history within past 6 months from the baseline

Exclusion Criteria:

* Diagnostic evidence of probable Alzheimer's disease consistent with National Institute of Neurological and Communicative Diseases and Stroke-Alzheimer's Disease and Related Disorders Association
* CDR-Global score (CDR-GS) >1
* Participant who has taken memantine, acetylcholinesterase inhibitors, or nootropics prior to participating in this study
* Any significant neurologic disease: other than suspected incipient Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
* Neuroimaging: participant with severe subcortical hyperintensities: D3-P3
* Magnetic resonance imaging exclusions: presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body
* Participant who is pregnant, lactating or of childbearing potential (i.e., women must be two years post-menopausal or surgically sterile)

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Rate of Alzheimer's Disease (AD) conversion differences between high-risk mild cognitive impairment (MCI) and low-risk MCI | Up to 36 months
  AD conversion differences will be assessed according to National Institute of Neurological and Communicative Diseases and Stroke-Alzheimer's Disease and Related Disorders Association Criteria for Probable AD.

SECONDARY OUTCOMES:
Mean change from Baseline in Seoul Neuropsychological Screening Battery-Dementia Version scores | Baseline, Month 12, Month 24
Mean change from Baseline in Clinical Dementia Rating (CDR) Sum of Boxes scores | Baseline, Month 12, Month 24
Mean change from Baseline in the CDR-Global Score | Baseline, Month 12, Month 24
Mean change from Baseline in Geriatric Depression Scale scores | Baseline, Month 12, Month 24
Mean change from Baseline in the volume of the whole brain according to Baseline demographics | Baseline, Month 12, Month 24
Mean change from Baseline in other structural magnetic resonance imaging (MRI) measures according to Baseline demographics | Baseline, Month 12, Month 24
Mean change from Baseline in the volume of the hippocampus according to Baseline demographics | Baseline, Month 12, Month 24

CONTACTS AND LOCATIONS:
Locations (16):
- South Korea (16):
  - Eisai Trial site_12, Anyang
  - Eisai Trial site_11, Busan
  - Eisai Trial site_15, Busan
  - Eisai Trial site_08, Changwon
  - Eisai Trial site_09, Daegu
  - Eisai Trial site_05, Daejeon
  - Eisai Trial site_03, Gachon
  - Eisai Trial site_07, Guri-si
  - Eisai Trial site_10, Gwangju
  - Eisai Trial site_16, Jeju City
  - Eisai Trial site_01, Seoul
  - Eisai Trial site_02, Seoul
  - Eisai Trial site_04, Seoul
  - Eisai Trial site_06, Seoul
  - Eisai Trial site_13, Seoul
  - Eisai Trial site_14, Seoul

REFERENCES:
- [Derived] Jang H, Na DL, Kwon JC, Jung NY, Moon Y, Lee JS, Park KW, Lee AY, Cho H, Lee JH, Kim BC, Park KH, Lee BC, Choi H, Kim J, Park MY. A Two-Year Observational Study to Evaluate Conversion Rates from High- and Low-Risk Patients with Amnestic Mild Cognitive Impairment to Probable Alzheimer's Disease in a Real-World Setting. J Alzheimers Dis Rep. 2024 May 17;8(1):851-862. doi: 10.3233/ADR-230189. eCollection 2024. PMID 38910942